CLINICAL TRIAL: NCT07132125
Title: Conversations With AI Chatbots Increase Short-Term Vaccine Intentions But Do Not Outperform Standard Public Health Messaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LLM_857299
Record Dates: First submitted 2025-08-12; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: HPV Vaccination Intent
Keywords: chatbot; artificial intelligence; large language models; HPV vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Default-style LLM chatbot (Experimental): A large language model chatbot (GPT-4o) that delivers tailored persuasive messages to parents about HPV vaccination, using the model's default style with longer, structured responses. Participants engage in a three-minute, multi-turn conversation, with responses personalized to their top-rated vaccine concern identified in a pre-intervention survey.
  Interventions: Behavioral: Default-style LLM chatbot
- Conversational-style LLM chatbot (Experimental): A large language model chatbot (GPT-4o) that delivers tailored persuasive messages to parents about HPV vaccination in a conversational style, with short responses. Participants engage in a three-minute, multi-turn conversation, with responses personalized to their top-rated vaccine concern identified in a pre-intervention survey.
  Interventions: Behavioral: Conversational-style LLM chatbot
- Public health informational materials (Active Comparator): Official public health informational materials on HPV vaccination from the Centers for Disease Control and Prevention (U.S.), National Health Service (U.K.), or Public Health Agency of Canada, matched to the participant's country of residence. Materials are 589-680 words in length, cover HPV risks and benefits of vaccination, and are presented for three minutes before participants proceed.
  Interventions: Behavioral: Public health informational materials
- No Message (No Intervention): No Intervention

INTERVENTIONS:
Behavioral: Default-style LLM chatbot — A large language model chatbot (GPT-4o) that delivers tailored persuasive messages to parents about HPV vaccination, using the model's default style with longer, structured responses. Participants engage in a three-minute, multi-turn conversation, with responses personalized to their top-rated vaccine concern identified in a pre-intervention survey.
  Arms: Default-style LLM chatbot
Behavioral: Conversational-style LLM chatbot — A large language model chatbot (GPT-4o) that delivers tailored persuasive messages to parents about HPV vaccination in a conversational style, with short responses. Participants engage in a three-minute, multi-turn conversation, with responses personalized to their top-rated vaccine concern identified in a pre-intervention survey.
  Arms: Conversational-style LLM chatbot
Behavioral: Public health informational materials — Official public health informational materials on HPV vaccination from the Centers for Disease Control and Prevention (U.S.), National Health Service (U.K.), or Public Health Agency of Canada, matched to the participant's country of residence. Materials are 589-680 words in length, cover HPV risks and benefits of vaccination, and are presented for three minutes before participants proceed.
  Arms: Public health informational materials

SUMMARY:
The goal of this clinical trial is to test whether short conversations with large language model (LLM) chatbots can persuade vaccine-hesitant parents to vaccinate their children against human papillomavirus (HPV). The study compares two chatbot styles to official public health information and to a no-message control. Parents of HPV-eligible children first complete a survey about their attitudes toward the HPV vaccine and their main concerns. They are then randomly assigned to read public health materials, have a three-minute conversation with either a default-style chatbot or a conversational-style chatbot tailored to their concern, or receive no message. The main outcome is change in intent to vaccinate immediately after the intervention, with follow-up surveys at 15 and 45 days.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and up
* Living in Canada, the UK, or the USA
* At least one child eligible for HPV vaccine based on country-specific guidelines who has not received any doses of the vaccine or whose vaccination status is unknown

Exclusion Criteria:

* Failure to pass attention checks
* Identified as non-human respondents by reCAPTCHA or other automated bot detection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 930 (Actual)
Dates: Start 2025-03-17 (Actual); Primary Completion 2025-05-22 (Actual); Study Completion 2025-05-22 (Actual)

PRIMARY OUTCOMES:
Change in intent to vaccinate child against HPV within the next 12 months | Baseline to immediately post-intervention
  Self-reported likelihood, on a 0-100 scale, of vaccinating the participant's youngest HPV vaccine-eligible child (identified in pre-survey) within the next 12 months. Measured before and immediately after the intervention to assess short-term changes in vaccination intent.

SECONDARY OUTCOMES:
Change in intent to vaccinate child against HPV at 15-day follow-up | Baseline to 15 days post-intervention
  Self-reported likelihood, on a 0-100 scale, of vaccinating the participant's youngest HPV vaccine-eligible child within the next 12 months. Measured at baseline and 15 days after the intervention to assess durability of effects.
Change in intent to vaccinate child against HPV at 45-day follow-up | Baseline to 45 days post-intervention
  Self-reported likelihood, on a 0-100 scale, of vaccinating the participant's youngest HPV vaccine-eligible child within the next 12 months. Measured at baseline and 45 days after the intervention to assess durability of effects.
Change in general parental vaccine hesitancy (PACV-5) | Baseline to immediately post-intervention
  Change in scores on the 5-item Parent Attitudes about Childhood Vaccines (PACV-5) scale. Measured at baseline and immediately after the intervention.
Change in intent to vaccinate child for influenza and COVID-19 | Measured at baseline and immediately post-intervention.
  Self-reported likelihood, on a 0-100 scale, of vaccinating the participant's youngest eligible child for influenza or COVID-19 within the next 12 months.
Change in importance ratings of HPV vaccine concerns | Baseline to immediately post-intervention
  Change in participant ratings (0-100 scale) of importance for each HPV vaccine concern (list derived from National Immunization Surveys) between baseline and immediately post-intervention.
Clicks on HPV vaccine appointment scheduling link | Immediately post-intervention
  Whether participants click a provided link to schedule an HPV vaccine appointment through CVS during the post-intervention survey.
Willingness to donate payment to vaccine education charity | Immediately post-intervention
  Percentage of survey payment participants choose to donate (0%, 10%, 30%, or 50%) to an immunization-related charity during the post-intervention survey.
Willingness to be recontacted for future research | Immediately post-intervention
  Participant self-reported willingness (yes/no) to be contacted for future studies
Ratings of empathy, usefulness, and relevance of intervention content | Immediately post-intervention
  Participant ratings (1-5 scale) of how empathetic, useful, and relevant they found the assigned chatbot conversation or public health reading material.

CONTACTS AND LOCATIONS:
Locations (1):
- Participants are recruited online via Prolific, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes